CLINICAL TRIAL: NCT02133066
Title: The Effect of Bedside Ultrasound Assistance on the Proportion of Successful Infant Lumbar Punctures in a Pediatric Emergency Department: A Randomized Controlled Trial
Brief Title: The Effect of Bedside Ultrasound Assistance on the Proportion of Successful Infant Spinal Taps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-010667
Record Dates: First submitted 2014-05-02; First posted 2014-05-07 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Traumatic Lumbar Puncture
Keywords: Ultrasound; Lumbar Puncture; Spinal Tap; Pediatric; Infant; Bedside Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- US-Assisted site marking for Lumbar Punctures (LP) (Active Comparator): Mindray M7 Ultrasound marking
  Interventions: Procedure: Bedside Ultrasound-Assisted Site Marking; Device: Mindray M7 Ultrasound
- Routine lumbar puncture (Placebo Comparator): These patients will receive no ultrasound-assisted site marking prior to lumbar puncture; The patients will simply have a "standard-of-care" spinal tap performed by the clinician
  Interventions: Procedure: Routine lumbar puncture

INTERVENTIONS:
Procedure: Bedside Ultrasound-Assisted Site Marking — Patient will receive a bedside ultrasound-assisted site marking of the most appropriate site for lumbar puncture prior to the clinician completing the spinal tap using Mindray M7 Ultrasound.
  Other Names: Mindray M7 Ultrasound
  Arms: US-Assisted site marking for Lumbar Punctures (LP)
Device: Mindray M7 Ultrasound — Patient will receive a bedside ultrasound exam of the most appropriate site for lumbar puncture prior to the clinician completing the spinal tap
  Other Names: M7/M7T Diagnostic Ultrasound
  Arms: US-Assisted site marking for Lumbar Punctures (LP)
Procedure: Routine lumbar puncture — Lumbar puncture will be performed per routine standard of care
  Arms: Routine lumbar puncture

SUMMARY:
The reported rate of unsuccessful spinal taps in children, especially young infants, is high. Our hypothesis is that ultrasound assistance can improve the success rate of spinal taps.

DETAILED DESCRIPTION:
The reported rate of unsuccessful spinal taps in children is high. At the Children's Hospital of Philadelphia (CHOP), quality improvement data demonstrates a failure rate of ~40-50%. Research has shown that bedside ultrasound can improve visualization and improve the success rate of spinal taps. Increasing the proportion of successful spinal taps in the emergency department could significantly reduce the rate of unnecessary hospitalizations, additional interventional procedures and antibiotic use. Our objective is to determine if bedside ultrasound-assisted site marking will increase the proportion of first attempt successful spinal taps. This will be a prospective, randomized controlled study that will take place over the course of 18 months with the goal to recruit a sample of approximately 128 patients. We will recruit subjects from the CHOP Emergency Department. The patients will be randomized into an ultrasound-assisted group versus a non-ultrasound-assisted group. Our hypothesis is that bedside ultrasound-assisted site marking will increase the number of successful spinal taps.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to six months of age
* Plan for diagnostic or therapeutic lumbar puncture as per front line clinician
* Availability of a study sonographer to perform bedside ultrasound

Exclusion Criteria:

* Known spinal cord abnormality (e.g., tethered cord, spina bifida)

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Chen, MD, Principal Investigator — CHOP
Locations (1):
- Children's Hospital of Philadelphia Emergency Department, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Abo A, Chen L, Johnston P, Santucci K. Positioning for lumbar puncture in children evaluated by bedside ultrasound. Pediatrics. 2010 May;125(5):e1149-53. doi: 10.1542/peds.2009-0646. Epub 2010 Apr 19. PMID 20403933
- [Background] Baxter AL, Fisher RG, Burke BL, Goldblatt SS, Isaacman DJ, Lawson ML. Local anesthetic and stylet styles: factors associated with resident lumbar puncture success. Pediatrics. 2006 Mar;117(3):876-81. doi: 10.1542/peds.2005-0519. PMID 16510670
- [Background] Bruccoleri RE, Chen L. Needle-entry angle for lumbar puncture in children as determined by using ultrasonography. Pediatrics. 2011 Apr;127(4):e921-6. doi: 10.1542/peds.2010-2511. Epub 2011 Mar 28. PMID 21444601
- [Background] Coley BD, Murakami JW, Koch BL, Shiels WE 2nd, Bates G, Hogan M. Diagnostic and interventional ultrasound of the pediatric spine. Pediatr Radiol. 2001 Nov;31(11):775-85. doi: 10.1007/s002470100535. PMID 11692234
- [Background] Dietrich AM, Coley BD. Bedside pediatric emergency evaluation through ultrasonography. Pediatr Radiol. 2008 Nov;38 Suppl 4:S679-84. doi: 10.1007/s00247-008-0890-1. Epub 2008 Sep 23. PMID 18810417
- [Background] Ferre RM, Sweeney TW. Emergency physicians can easily obtain ultrasound images of anatomical landmarks relevant to lumbar puncture. Am J Emerg Med. 2007 Mar;25(3):291-6. doi: 10.1016/j.ajem.2006.08.013. PMID 17349903
- [Background] Furness G, Reilly MP, Kuchi S. An evaluation of ultrasound imaging for identification of lumbar intervertebral level. Anaesthesia. 2002 Mar;57(3):277-80. doi: 10.1046/j.1365-2044.2002.2403_4.x. PMID 11892638
- [Background] Lam WW, Ai V, Wong V, Lui WM, Chan FL, Leong L. Ultrasound measurement of lumbosacral spine in children. Pediatr Neurol. 2004 Feb;30(2):115-21. doi: 10.1016/j.pediatrneurol.2003.07.002. PMID 14984904
- [Background] Nigrovic LE, Kuppermann N, Neuman MI. Risk factors for traumatic or unsuccessful lumbar punctures in children. Ann Emerg Med. 2007 Jun;49(6):762-71. doi: 10.1016/j.annemergmed.2006.10.018. Epub 2007 Feb 23. PMID 17321005
- [Background] Nigrovic LE, Shah SS, Neuman MI. Correction of cerebrospinal fluid protein for the presence of red blood cells in children with a traumatic lumbar puncture. J Pediatr. 2011 Jul;159(1):158-9. doi: 10.1016/j.jpeds.2011.02.038. Epub 2011 Apr 14. PMID 21492866
- [Background] Nomura JT, Leech SJ, Shenbagamurthi S, Sierzenski PR, O'Connor RE, Bollinger M, Humphrey M, Gukhool JA. A randomized controlled trial of ultrasound-assisted lumbar puncture. J Ultrasound Med. 2007 Oct;26(10):1341-8. doi: 10.7863/jum.2007.26.10.1341. PMID 17901137
- [Background] Oncel S, Gunlemez A, Anik Y, Alvur M. Positioning of infants in the neonatal intensive care unit for lumbar puncture as determined by bedside ultrasonography. Arch Dis Child Fetal Neonatal Ed. 2013 Mar;98(2):F133-5. doi: 10.1136/archdischild-2011-301475. Epub 2012 Jun 9. PMID 22684159
- [Background] Pappano D. "Traumatic tap" proportion in pediatric lumbar puncture. Pediatr Emerg Care. 2010 Jul;26(7):487-9. doi: 10.1097/PEC.0b013e3181e5bedd. PMID 20577138
- [Background] Peterson MA, Abele J. Bedside ultrasound for difficult lumbar puncture. J Emerg Med. 2005 Feb;28(2):197-200. doi: 10.1016/j.jemermed.2004.09.008. PMID 15707816
- [Background] Pinheiro JM, Furdon S, Ochoa LF. Role of local anesthesia during lumbar puncture in neonates. Pediatrics. 1993 Feb;91(2):379-82. PMID 8424014
- [Background] Schreiner RL, Kleiman MB. Incidence and effect of traumatic lumbar puncture in the neonate. Dev Med Child Neurol. 1979 Aug;21(4):483-7. doi: 10.1111/j.1469-8749.1979.tb01652.x. PMID 520695
- [Background] Srinivasan L, Shah SS, Abbasi S, Padula MA, Harris MC. Traumatic lumbar punctures in infants hospitalized in the neonatal intensive care unit. Pediatr Infect Dis J. 2013 Oct;32(10):1150-2. doi: 10.1097/INF.0b013e31829862b7. PMID 23624433

RESULTS

PARTICIPANT FLOW:
Groups:
- US-Assisted Site Marking for LP: Mindray M7 Ultrasound marking
  Bedside Ultrasound-Assisted Site Marking: Patient will receive a bedside ultrasound-assisted site marking of the most appropriate site for lumbar puncture prior to the clinician completing the spinal tap using Mindray M7 Ultrasound.
  Mindray M7 Ultrasound: Patient will receive a bedside ultrasound exam of the most appropriate site for lumbar puncture prior to the clinician completing the spinal tap
Period: Overall Study
Arm/Group | US-Assisted Site Marking for LP | Routine Lumbar Puncture
Started | 64 | 64
Completed | 64 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | US-Assisted Site Marking for LP | Routine Lumbar Puncture | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 64 | 128
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: days] | 24 [9 to 34] | 29 [14 to 45] | 26 [3 to 179]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 34 | 53
  Male | 45 | 30 | 75
Region of Enrollment [Number; unit: participants]
  United States | 64 | 64 | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful First Attempt Lumbar Punctures in the Ultrasound-assisted Group as Compared to the Non-ultrasound Assisted Group
Description: First attempt success in ultrasound-assisted group compared to first attempt success in non-ultrasound assisted group
Time Frame: 30 minutes
Measure: Number (95% Confidence Interval); unit: percent success
Arm/Group | US-Assisted Site Marking for LP | Routine Lumbar Puncture
Number analyzed (Participants) | 64 | 64
percent success | 58 [50 to 70] | 31 [19 to 39]

2. Secondary Outcome: Percentage of Overall Success of Lumbar Punctures in the Ultrasound-assisted Group Versus the Non-ultrasound-assisted Group
Description: Overall success of lumbar punctures (within 3 attempts) in the non-ultrasound-assisted group compared to the ultrasound-assisted group
Time Frame: 30 minutes
Measure: Number (95% Confidence Interval); unit: percentage success
Arm/Group | US-Assisted Site Marking for LP | Routine Lumbar Puncture
Number analyzed (Participants) | 64 | 64
percentage success | 75 [68 to 82] | 44 [38 to 52]

3. Secondary Outcome: Length of Hospitalization in Ultrasound-assisted Lumbar Puncture Patients Versus Non-ultrasound-assisted Patients
Description: If a lumbar puncture is not successful, this may lead to a longer hospitalization than necessary until a lumbar puncture can be completed (with interventional radiology or other resources). According to our hypothesis, we believe that ultrasound assistance will increase the proportion of successful lumbar punctures, and therefore, decrease the length of unnecessary hospitalization.
Time Frame: Participants will be followed for the duration of the hospital stay, an expected average of 2 days
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | US-Assisted Site Marking for LP | Routine Lumbar Puncture
Number analyzed (Participants) | 64 | 64
hours | 46 [35 to 61] | 48.1 [37 to 62]

4. Secondary Outcome: Length of Antibiotic Use in Ultrasound-assisted Lumbar Puncture Patients Versus Non-ultrasound-assisted Patients
Description: If a lumbar puncture is not successful, this may lead to unnecessary (prophylactic) antibiotic use until a lumbar puncture can be completed (with interventional radiology or other resources) to rule out meningitis. According to our hypothesis, we believe that ultrasound assistance will increase the proportion of successful lumbar punctures, and therefore, decrease the length of unnecessary antibiotics.
Time Frame: Participants will be followed until discontinuation of antibiotics, an expected average of 2 days
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | US-Assisted Site Marking for LP | Routine Lumbar Puncture
Number analyzed (Participants) | 64 | 64
hours | 26.8 [19 to 30] | 25 [18 to 29]

ADVERSE EVENTS:
Arm/Group | US-Assisted Site Marking for LP | Routine Lumbar Puncture
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes